CLINICAL TRIAL: NCT02188888
Title: Heart Rate Reduction With Esmolol is Associated With Improved Arterial Elastance in Patients With Septic Shock. A Prospective Observational Study
Brief Title: Echocardiographic and Arterial Pressure Waveform Changes After Reducing Heart Rate With Esmolol in Septic Shock Patients
Status: Completed | Type: Observational
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Andrea Morelli, associate professor, University of Roma La Sapienza
Other Study IDs: 2309
Record Dates: First submitted 2014-07-10; First posted 2014-07-14 (Estimated); Last update posted 2015-08-07 (Estimated); Status verified 2015-08

CONDITIONS: Tachycardia; Septic Shock
Keywords: septic shock; esmolol; tachycardia; betablockers
MeSH Terms: conditions — Tachycardia; Shock, Septic | interventions — esmolol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Tachycardic patients: Patients will receive a continuous esmolol infusion to maintain heart rate between 94 and 80 bpm. Norepinephrine will be titrated to achieve a MAP between 65 and 75 mmHg.
  Interventions: Drug: esmolol

INTERVENTIONS:
Drug: esmolol — Strict heart rate control: esmolol at any dose to maintain heart rate between 95 and 80 bpm

SUMMARY:
Clinical study suggests that beta-blockers by decreasing heart rate together with an increase in stroke volume do not negatively affect cardiac output allowing an economization of cardiac work and oxygen consumption in patients with septic shock. Whether this hemodynamic profile leads to an amelioration of myocardial performance is still unclear. The objective of the present study is therefore to elucidate whether a reduction in heart rate with esmolol is associated to an improvement of cardiac efficiency in patients with septic shock who remained tachycardic after hemodynamic optimization.

DETAILED DESCRIPTION:
After 24-36 hours of initial hemodynamic stabilization, 44 septic shock patients with heart rate > of 95 bpm and requiring norepinephrine to maintain mean arterial pressure (MAP) between 65 and 75 mmHg despite adequate volume resuscitation,will receive a continuous esmolol infusion to maintain heart rate between 94 and 80 bpm. Norepinephrine will be titrated to achieve a MAP between 65 and 75 mmHg. To investigate myocardial performance, we will simultaneously assess LV ejection fraction (LVEF), tricuspidal annular plane solid excursion (TAPSE) by echocardiography, the dP/dt MAX and the cardiac cycle efficiency (CCE) both estimated from the arterial pressure waveform. Finally we will analyze changes in static arterial elastance. Data will be obtained at baseline and after four hours once achieved the predefined heart rate threshold.

ELIGIBILITY:
Inclusion Criteria:

* septic shock criteria
* presence of heart rate > 95 bpm.

Exclusion Criteria:

* Pregnancy
* age < 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Septic shock patients with heart rate > of 95 bpm and requiring norepinephrine to maintain mean arterial pressure (MAP) between 65 and 75 mmHg after at least 24 hours of hemodynamic optimization.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2013-12; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
heart rate | over a period of four hours

SECONDARY OUTCOMES:
echocardiography | over a period of four hours
  LV ejection fraction (LVEF) and tricuspidal annular plane solid excursion (TAPSE)
static arterial elastance | over a period of four hours

OTHER OUTCOMES:
arterial pressure waveform | over a period of four hours
  systolic, diastolic and dicrotic pressures

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Morelli, MD, Principal Investigator — University of Roma La Sapienza
Locations (1):
- Department of Anesthesiology and Intensive care of the University of Rome La Sapienza, Rome, Italy

REFERENCES:
- [Derived] Morelli A, Romano SM, Sanfilippo F, Santonocito C, Frati G, Chiostri M, Agro FE, Ertmer C, Rehberg SW, Vieillard-Baron A. Systolic-dicrotic notch pressure difference can identify tachycardic patients with septic shock at risk of cardiovascular decompensation following pharmacological heart rate reduction. Br J Anaesth. 2020 Dec;125(6):1018-1024. doi: 10.1016/j.bja.2020.05.058. Epub 2020 Jul 18. PMID 32690246